CLINICAL TRIAL: NCT00263341
Title: A Multicenter, Open-label Study on the Efficacy, Cycle Control and Safety of a Contraceptive Vaginal Ring Delivering a Daily Dose of 150 ug of Nestorone® and 15 ug of Ethinyl Estradiol
Brief Title: Safety and Efficacy of a Contraceptive Vaginal Ring Delivering Nestorone® and Ethinyl Estradiol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Protocol 300
Record Dates: First submitted 2005-12-06; First posted 2005-12-08 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Contraception
Keywords: Contraceptive agents; Female contraception; Progestins
MeSH Terms: interventions — ST 1435; segesterone acetate and ethinyl estradiol vaginal system

INTERVENTIONS:
Combination Product: NES/EE CVR — This is a Phase 3, multicenter, open-label study of a 21/7-day regimen of the 150/15 NES/EE CVR, in healthy women followed on an outpatient basis up to one year (13 cycles) of treatment over one year. Because of the stop treatment date of December 31, 2008 for all participants, women enrolling or re-enrolling in 2008 may not complete a full 13 cycles of treatment. Subjects may also participate in a 6 month follow-up period after the 300B study. The ring is designed to last for 12 months.
  Other Names: Nestorone (segesterone acetate) Ethinylestradiol Contraceptive Vaginal Ring

SUMMARY:
The purpose of this 1-year study is to evaluate the efficacy and safety of a new contraceptive vaginal ring (CVR) delivering low doses of Nestorone (NES), a new, nonandrogenic progestin, and ethinyl estradiol (EE), an estrogen used in oral contraceptives. The CVR, which is made of silicone rubber, is designed to be used for 1 year (13 menstrual cycles) before replacement is required.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the contraceptive efficacy, cycle control, and safety of a reusable CVR delivering low daily doses of NES and EE for a 1-year (13-cycle) period.

Nestorone is a potent, nonandrogenic, 19-norprogesterone derivative, which is not active when given orally, but is highly active when delivered via non-oral delivery systems, such as CVRs, implants, or transdermal preparations. The high potency of NES makes it an excellent candidate for use in contraceptive delivery systems designed to be effective for prolonged periods. This characteristic of Nestorone has been utilized in the design of a contraceptive vaginal ring that releases low daily doses of both NES and EE and is effective for a 1-year (13-cycle) period. The NES/EE vaginal ring is a long-acting contraceptive device, but, unlike other long-term methods, it use is controlled by the woman without the need for medical intervention.

The efficacy of NES/EE vaginal ring in preventing pregnancy during a 1-year (13-cycle) period will be studied in women who have regular sexual activity and use no other form of contraception. The Pearl index for all women (18-<40) and Kaplan-Meier life table analyses will be assessed for all subjects and for subjects £ 35 years and will provide supportive analyses for demonstrating efficacy. Pearl indices will be based on all cycles and on all cycles for which back-up contraception is not used.

The number of bleeding/spotting days per cycle or reference period will be used to evaluate cycle control. Safety will be evaluated by regular assessments of blood pressure, pulse, and body weight and by laboratory testing and Pap smears at screening and termination, and by the frequencies of adverse events and serious adverse events. Additional safety evaluations will be obtained in a companion Phase 3 study conducted by the NIH (Protocol CCN006) with three substudies to evaluate 1) the effect of treatment on 4 hepatic proteins that may be associated with a risk for thromboembolism; 2) the effect of reusing the same CVR for 13 consecutive cycles on vaginal flora and the risk of infection; and 3) the effect of vaginal delivery of NES and EE on the endometrium.

A nested pharmacokinetics/pharmacodynamics/safety study is also being conducted in a subset of 39 patients. Blood samples are drawn during study cycles 1, 3, and 13 in order to assess ovulation suppression, measured by serum progesterone concentration, and the pharmacokinetics of NES and EE.

ELIGIBILITY:
Inclusion Criteria:

Healthy women who meet the following criteria:

* Aged 18-<40 years who wish to use a combined hormonal contraceptive.
* Women not intending to become pregnant for 13 months.
* Intact uterus and both ovaries.
* Prior history of regular menstrual cycles of 28 ± 7 days when not using hormonal contraception; if postpartum or postabortal, history of regular menstrual cycles of 21-35 days in length and at least one cycle (2 menses) with a cycle length consistent with her past cycles.
* Sexually active (currently) and willing to discontinue current contraceptive method to participate in the study.
* In the opinion of the investigator, able to comply with the protocol, e.g. live within the clinic catchment area or within a reasonable distance from the clinic.
* Do not meet any of the exclusion criteria.
* Signed informed consent prior to entry into the trial.

[For pharmacokinetics study only; 39 subjects already recruited]

- Willing to undergo frequent blooding sampling

Exclusion Criteria:

Contraindications for enrollment will be the same as those for use with combined hormonal contraceptives in addition to contraindications specific to this clinical trial including:

* Known hypersensitivity to estrogens or progestins.
* Known hypersensitivity to silicone rubber.
* Known or suspected pregnancy.
* History of infertility of >1.0 year in woman or her male partner.
* History of vasectomy or sterility in male partner; tubal ligation (sterilization) in women.
* Undiagnosed abnormal genital bleeding.
* Undiagnosed vaginal discharge or vaginal lesions or abnormalities. (Subjects diagnosed at screening with a chlamydia or gonococcus infection may be included in the trial following treatment; partner treatment is also recommended. Investigators should make a determination if subjects are at high risk for reinfection, e.g. multiple sex partners, untreated partner, and whether such subjects can be included.)
* History of pelvic inflammatory disease since last pregnancy episode.
* History of toxic shock syndrome.
* Current abnormal Pap smear (women who have abnormal Paps but are ASCUS HPV negative may participate provided there is follow up for this finding per standard of care).
* Cystoceles or rectoceles or other anatomical abnormality that would preclude use of a vaginal ring.
* Women planning to undergo major surgery.
* Smoking in women who are 35 years and over or will be 35 years during the course of the trial; women < 35yrs who smoke 15 cigarettes or more must be evaluated by the PI for inclusion based on risk factors that would increase their risk for CVD, e.g. lipid levels, glucose level, BP, BMI, family history of CVD at a young age.
* Breastfeeding.
* Current or past thrombophlebitis or thromboembolic disorders.
* History of venous thrombosis or embolism in a first-degree relative, <55 years of age suggesting a familial defect in the blood coagulation system, which in the opinion of the PI, suggests use of a hormonal contraceptive could pose a significant risk.
* Cerebrovascular or cardiovascular disease.
* History of retinal vascular lesions, unexplained partial or complete loss of vision.
* Known or suspected carcinoma of the breast.
* Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia.
* Past history of any other carcinoma unless in remission for more than 5 years.
* Current or history of medically diagnosed severe depression, which, in the opinions of the investigator, could be exacerbated by use of a hormonal contraceptive.
* Headaches with focal neurological symptoms.
* Severe constipation.
* History of cholestatic jaundice of pregnancy or jaundice with prior steroid use.
* Benign or malignant liver tumors; active liver disease.
* Diastolic blood pressure (BP) 85 mm Hg and/or systolic BP 135 mm Hg after 5-10 minutes rest.
* Known or suspected alcoholism or drug abuse.
* Abnormal serum chemistry values according to the physician's judgment.
* Participation in another clinical trial within last 30 days.
* Weight >95 kg or >209 lbs.
* Use of liver enzyme inducers on a regular basis.
* Use of monthly injectable contraceptives (e.g. cyclofem) unless suspended 2 months before initiation of treatment. Use of Depo-Provera [depo-medroxyprogesterone (DMPA)] unless suspended 6 months before treatment.
* Current use of implanted hormonal contraceptives, including Mirena® [progestin containing intrauterine system (IUS)], Jadelle®, Norplant® or Implanon® (subjects using any of these methods who request removal for reasons unrelated to the purpose of enrollment in this study may be considered for participation).
* Current use of a non-hormonal IUD. Subjects with IUDs who request removal for reasons unrelated to the purpose of enrollment in this study may be considered for participation.
* Known HIV infection.
* Women at high risk of contracting HIV, e.g. women with multiple sex partners who need to use condoms consistently, injection drug users. If women enrolled in the study do use condoms to protect against STIs, they should be instructed that this occasional use should be with non-N-9 containing condoms and they should record condom use in their diaries. Women found to have an STI at screening will be treated prior to inclusion in the study (with the exception of those infected with HIV).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1135 (Actual)
Dates: Start 2005-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Efficacy | At all visits
  Primary endpoint: The Pearl Index for women 35 years of age derived from using all cycles for which back up contraception is not used will be the primary efficacy endpoint. This index will be calculated for the women participating in Protocol 300 B and will then be pooled with data from women 35 years who participate in 300 A (CCN006).
Safety | At all visits
  Each subject's health status will be monitored carefully throughout the trial. Baseline data collected at the screening visit will consist of the medical and gynecologic history and physical examination findings including breast and pelvic exam (to include Pap test and STI screening for chlamydia and gonorrhea). These assessments will be repeated at the 6th cycle visit (with the exception of the Pap, and STI screening). Baseline data obtained from clinical chemistries and a CBC will be used to monitor liver and renal function, lipid levels and hematologic status.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Merkatz, Ph.D., Study Director — Population Council
Locations (12):
- United States (5):
  - Women and Children's Hospital, LAC/USC Medical Center, Los Angeles, California
  - University of California, San Francisco General Hospital, Department of Obstetrics & Gynecology, San Francisco, California
  - University of Chicago Hospitals, Chicago, Illinois
  - Montefiore Medical Center/Albert Einstein College of Medicine, The Bronx, New York
  - Columbus Center for Women's Heatlh Research, Columbus, Ohio
- FPA Health, Ashfield, Australia
- University of Campinas, Department of Obstetrics & Gynecology, São Paulo, Brazil
- Instituto Chileno de Medicina Reproductiva, Santiago, Chile
- Profamilia, Santo Domingo, Dominican Republic
- Family Federation of Finland, Helsinki, Finland
- University of Szeged, Department of Obstetrics & Gynecology, Szeged, Hungary
- Karolinska Institutet, Department of Woman and Child Health, Division of Obstetrics & Gynecology, Stockholm, Sweden

REFERENCES:
- [Derived] Plagianos MG, Ramanadhan S, Merkatz RB, Brache V, Friedland BA, Haddad LB. Risk factors for and outcomes of ring expulsions with a 1-year contraceptive vaginal system. Am J Obstet Gynecol. 2024 May;230(5):548.e1-548.e8. doi: 10.1016/j.ajog.2024.01.020. Epub 2024 Jan 29. PMID 38295968
- [Derived] Jensen JT, Archer DF, Westhoff CL, Nelson AL, Graham S, Bernick B. Satisfaction with a Segesterone Acetate and Ethinyl Estradiol Contraceptive Vaginal System Among Recent Oral Contraceptive or Hormonal Contraceptive Vaginal Ring Users. J Womens Health (Larchmt). 2023 Jul;32(7):808-815. doi: 10.1089/jwh.2022.0264. Epub 2023 May 29. PMID 37253139
- [Derived] Vieira CS, Fraser IS, Plagianos MG, Burke AE, Westhoff CL, Jensen J, Brache V, Bahamondes L, Merkatz R, Sitruk-Ware R, Blithe DL. Bleeding profile associated with 1-year use of the segesterone acetate/ethinyl estradiol contraceptive vaginal system: pooled analysis from Phase 3 trials. Contraception. 2019 Dec;100(6):438-444. doi: 10.1016/j.contraception.2019.07.145. Epub 2019 Aug 6. PMID 31398307
- [Derived] Archer DF, Merkatz RB, Bahamondes L, Westhoff CL, Darney P, Apter D, Jensen JT, Brache V, Nelson AL, Banks E, Bartfai G, Portman DJ, Plagianos M, Dart C, Kumar N, Creasy GW, Sitruk-Ware R, Blithe DL. Efficacy of the 1-year (13-cycle) segesterone acetate and ethinylestradiol contraceptive vaginal system: results of two multicentre, open-label, single-arm, phase 3 trials. Lancet Glob Health. 2019 Aug;7(8):e1054-e1064. doi: 10.1016/S2214-109X(19)30265-7. Epub 2019 Jun 20. PMID 31231065
- [Derived] Stifani BM, Plagianos M, Vieira CS, Merkatz RB. Factors associated with nonadherence to instructions for using the Nestorone(R)/ethinyl estradiol contraceptive vaginal ring. Contraception. 2018 May;97(5):415-421. doi: 10.1016/j.contraception.2017.12.011. Epub 2017 Dec 18. PMID 29269252
- [Derived] Huang Y, Merkatz RB, Hillier SL, Roberts K, Blithe DL, Sitruk-Ware R, Creinin MD. Effects of a One Year Reusable Contraceptive Vaginal Ring on Vaginal Microflora and the Risk of Vaginal Infection: An Open-Label Prospective Evaluation. PLoS One. 2015 Aug 12;10(8):e0134460. doi: 10.1371/journal.pone.0134460. eCollection 2015. PMID 26267119
- [Derived] Merkatz RB, Plagianos M, Hoskin E, Cooney M, Hewett PC, Mensch BS. Acceptability of the Nestorone(R)/ethinyl estradiol contraceptive vaginal ring: development of a model; implications for introduction. Contraception. 2014 Nov;90(5):514-21. doi: 10.1016/j.contraception.2014.05.015. Epub 2014 Jun 2. PMID 24993487